CLINICAL TRIAL: NCT06885775
Title: A Multicenter, Randomized, Evaluator- and Subject-blinded, Active-controlled, Paired, Confirmatory Clinical Trial to Compare and Evaluate the Efficacy and Safety of DXP01 Versus Juvéderm® ULTRA 3 in Adults Requiring the Temporary Improvement of Moderate to Severe Nasolabial Folds
Brief Title: Purpose of This Study is the Demonstration of Safety and Efficacy of the Dermal Fillers DXP01 Temporary Improvement of Moderate to Severe Nasolabial Folds
Acronym: DXP01
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: DEXLEVO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DXP01_NFE-01
Record Dates: First submitted 2025-02-20; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Dermal Fillers; Nasolabial Folds, Wrinkles
Keywords: NASOLABIAL FOLDS; DXP01

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participant, Investigator are blinded to treatment assignment to each side of their faces.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participant Group/Arm (Experimental): Device: DXP01 DXP01 is an opaque whit, containing polycaprolactone, carboxymethylcellulose, purified water in a injection solution, pre-filled in a syringe. Polycaprolactone is a 100% bioresorbable and highly biocompatible medical polymer that is metabolized and excreted through normal pathways as carbon dioxide (CO2) and water (H2O). Due to these properties, PCL fillers have received European CE certification and U.S. FDA approval as medical devices for dermal and subcutaneous insertion for wrinkle improvement since 2009.
  Interventions: Device: DXP01
- Treatment (Active Comparator): Device: Juvederm ULTRA 3 Description: Juvéderm® ULTRA 3 is a sterile pyrogen-free physiological solution of cross-linked hyaluronic (HA) acid which is not of animal origin. The gel is presented in a graduated, pre-filled, disposable syringe. Juvéderm® ULTRA 3 is an injectable implant used for filling mid and/ or deep depressions of the skin via mid and/or deep dermis injection, as well as for lip definition and enhancement.
  Interventions: Device: Juvederm ULTRA 3

INTERVENTIONS:
Device: DXP01 — PCL Dermal Filler
  Arms: Participant Group/Arm
Device: Juvederm ULTRA 3 — HA Dermal filler
  Arms: Treatment

SUMMARY:
Purpose of this study is the demonstration of safety and efficacy of the dermal fillers DXP01 Face for restoration of moderate to severe nasolabial folds

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational, two-arm, evaluator- and subject-blinded, active-controlled, paired clinical trial for demonstration of safety and efficacy of the dermal fillers DXP01 Face for restoration of moderate to severe nasolabial folds. Besides safety aspects, evaluated immediately after the treatment, 2 weeks, 8, 16, 24, 36 and 12 months after the treatment, the performance of the dermal fillers are evaluated in the 2, 8, 16, 24, 36 weeks and 12 months follow-up by using GAIS and WSRS.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 19 to 70 years.
2. Subjects with nasolabial folds (NLF) on both sides scored at 3 or 4 on the WSRS (Wrinkle Severity Rating Scale) as evaluated by the investigator at screening (both sides do not need to have the same score but must fall within the 3-4 range).
3. Subjects with visually symmetrical nasolabial folds (NLF) on both sides.
4. Subjects who can comply with the clinical trial procedures and will not undergo any facial cosmetic procedures/surgeries contraindicated for combination therapy during the clinical trial.
5. Males and females of childbearing potential who agree to use medically accepted contraception* during the clinical trial period. (*Hormonal contraception, intrauterine device (IUD) or intrauterine system (IUS), tubal ligation, double-barrier methods (such as combining cervical cap or diaphragm with male condom), or single-barrier methods combined with spermicide).
6. Subjects who have received a detailed explanation of this clinical trial, understand it, voluntarily decide to participate, and provide written consent.
7. For women of childbearing potential, individuals who test negative for pregnancy prior to the administration of the investigational product.

Exclusion Criteria:

1. Subjects with localized wounds or active infections (such as cysts, acne, rashes, hives, etc.) in the nasolabial fold area.
2. Subjects with acute, chronic, or recurrent skin conditions (whether infectious or non-infectious).
3. Subjects with scars or abnormal skin findings (such as moles, erythema, or telangiectasia) in the nasolabial fold area that may affect treatment outcomes.
4. Subjects with a history of keloid formation, hyperpigmentation, or hypertrophic scars.
5. Subjects with a history of bleeding disorders (such as liver disease, clotting factor deficiencies, etc.).
6. Subjects with a history of herpetic rash.
7. Subjects with connective tissue diseases, autoimmune diseases, or suspected immune deficiencies (such as Sjögren's syndrome, systemic lupus erythematosus, etc.).
8. Subjects with active sepsis, sarcoidosis, infective endocarditis, or confirmed infections regardless of location, type, or size.
9. Subjects with known allergies or hypersensitivity reactions, either localized or systemic, to the components of the investigational medical device or amide-type local anesthetics.
10. Subjects who tested positive in skin patch tests for either the investigational device or control device.
11. Subjects with a significant history of allergies or anaphylaxis that could affect this clinical trial.
12. Subjects with clinically significant disorders in the cardiovascular, gastrointestinal, respiratory, endocrine, or central nervous systems.
13. Subjects with a history of malignancy within 5 years of screening (except for those with basal cell carcinoma, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, thyroid cancer, or prostate cancer, provided there has been no recurrence for over 3 years after complete remission, as judged by the investigator).
14. Subjects suffering from untreated epilepsy.
15. Subjects suffering from porphyria.
16. Subjects with a history of alcohol or drug addiction.
17. Subjects with a history of psychiatric disorders that, in the investigator's opinion, could significantly affect this clinical trial.
18. Subjects who have undergone cosmetic procedures contraindicated for this clinical trial within 24 weeks of screening (except for upper eyelid surgery, rhinoplasty performed more than 24 months postoperatively, or lower eyelid correction).
19. Subjects who have undergone skin augmentation or permanent/semi-permanent implant-based cosmetic surgery (such as fillers based on CaHA, PLLA, PMMA, etc.) or PCL fillers or HA fillers on the face within 12 months of screening - CaHA (calcium hydroxyl apatite), PLLA (poly L-lactide), PMMA (polymethyl methacrylate), PCL (polycaprolactone), HA (Hyaluronic Acid)
20. Subjects who have taken any of the following medications within 1 week before the application of the investigational medical device or who are scheduled to take them within 3 days after application (however, if the medication is being taken at the time of screening and, in the investigator's judgment, a temporary discontinuation does not pose a medical risk, the individual may participate in the clinical trial after a 10-day wash-out period): *Anticoagulants, antiplatelet agents, thrombolytics (e.g., warfarin), oral/injectable corticosteroids, nonsteroidal anti-inflammatory drugs (NSAIDs) (low-dose aspirin up to 300 mg/day is permitted), and substances that delay blood coagulation time (such as vitamin E preparations of 400 IU/day or more, including multivitamins, garlic, and ginkgo biloba extracts).
21. Subjects who have received systemic corticosteroids or immune-suppressants within 12 weeks of screening.
22. Subjects who have applied oral or topical preparations or cosmetics with anti-wrinkle effects to the facial area within 12 weeks of screening (however, the use of sunscreen and certain cosmetics such as alpha hydroxyl acids, glycolic acids, retinol, or retinoic acids, which have been continuously used for more than 90 days prior to screening, is permitted).
23. Subjects who have undergone chemotherapy within 12 weeks of screening.
24. Subjects who have received botulinum toxin injections in the face within 24 weeks of screening.
25. Subjects who have taken other investigational drugs or had investigational medical devices applied within 4 weeks of screening.
26. Pregnant women, women planning to become pregnant during the clinical trial period, or breastfeeding women.
27. Subjects who, for any other reason, are deemed unsuitable by the investigator for inclusion in this clinical trial.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The difference in the WSRS (Wrinkle Severity Rating Scale) between the treatment groups at 24 weeks after device application, as evaluated by an independent assessor. | Baseline and week 24
  The primary objective of the study is to demonstrate the non-inferiority of DXP01 compared to Juvéderm® ULTRA 3 by assessing the mean WSRS (Wrinkle Severity Rating Scale) score at 24 weeks, as evaluated by an independent assessor, in adults with moderate to severe nasolabial folds after administration of DXP01 and Juvéderm® ULTRA 3.[The difference of WSRS(Wrinkle Severity Rating Scales) between baseline and week 24. A positive value indicated "effective" improvement; while a value of 0 or a negative value was regarded as "ineffective" treatment. And the WSRS improvement ratio was defined as the effective improvement ratio of either group.]

SECONDARY OUTCOMES:
• Efficacy of DXP01 as assessed by difference in the mean Wrinkle Severity Rating Scale (WSRS) score | • At 2, 8, 16, 36 and 48 weeks after device application
  • The mean value differences in the WSRS scores between group / The investigators calculated the mean value differences in the WSRS scores[Wrinkle severity assessment acc. to the Wrinkle Severity Rating Scale (WSRS); 1: wrinkles absent, 2: slight wrinkles, 3: moderate wrinkles, 4: severe wrinkles, 5: very severe wrinkles]
• Efficacy of DXP01 as assessed by difference in the mean Global Aesthetic Improvement Scale | • At 2, 8, 16, 36 and 48 weeks after device application
  • The mean value differences in the GAIS scores between group / The investigators calculated the mean value differences in the GAIS scores[GAIS: 3: very much improved, 2: much improved, 1: improved, 0 unchanged, -1: worse] between the test
• Product safety 2 weeks~48 weeks | • 2 weeks of treatment and during 48 weeks after treatment.
  • Short- and long-term adverse effects
• The mean value differences in the Pain Score Using Visual Analog Pain Scale(VAS) between | • After 15, 30, 45, 60 minutes(Immediate post-injection)
  • The VAS scale uses a 100 mm line labelled at '0' with 'no pain' and '100' with 'worst pain'.

CONTACTS AND LOCATIONS:
Locations (1):
- Societatea Civila Medicala Dr. Rosu, Romania, Timisoara, Romania